CLINICAL TRIAL: NCT03699735
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - Sonova2018_31
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_31
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Each participant will be treated with each test condition in a randomized order.
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hearing Aid with beam form principle_A (Active Comparator): Device: Hearing Aid beam former principle_A (simulation of real ear condition). Each participant will be fitted with the 3 different beam former (directionality change) principles on the same hearing aid, saved to 3 manual programs. Beam former principle is a sound processing algorithm to focus to a target source in a noisy situation to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of beam forming and good speech quality.
  Interventions: Device: Bolero B90-SP
- Hearing Aid with beam form principle_B (Experimental): Device: Hearing Aid beam former principle_B. Each participant will be fitted with the 3 different beam former (directionality change) principles on the same hearing aid, saved to 3 manual programs. Beam former principle is a sound processing algorithm to focus to a target source in a noisy situation to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of beam forming and good speech quality.
  Interventions: Device: Bolero B90-SP
- Hearing Aid with beam form principle_C (Experimental): Device: Hearing Aid beam former principle_C. Each participant will be fitted with the 3 different beam former (directionality change) principles on the same hearing aid, saved to 3 manual programs. Beam former principle is a sound processing algorithm to focus to a target source in a noisy situation to improve the speech intelligibility and comfort. The experimental conditions vary in their parametrization to result in different degrees of beam forming and good speech quality.
  Interventions: Device: Bolero B90-SP

INTERVENTIONS:
Device: Bolero B90-SP — Behind the ear Hearing device fitted with an individual ear mold to compensate a Hearing loss

SUMMARY:
A methodical evaluation of sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and asses strength and weaknesses of these sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Objective laboratory measurements will be carried out. This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with or without experience with hearing aids
* Sensorineural hearing loss (N4-N6 according to ISO 60118-15)
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Informed Consent as documented by signature
* Symmetric hearing loss below 1000 Hz

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments on study site
* Inability to produce a reliable hearing test result
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Individual binaural Hearing abilities | 2 weeks
  Primary Outcome measurement is to measure the speech understanding in noise [SNR in dB] for the beam former principles A, B and C

SECONDARY OUTCOMES:
Speechunderstanding for different beam form principles | 2 weeks
  Secondary Outcome measurement is to measure individual binaural Hearing abilities with psycho acoustical test principles (Binaural inter aural Level difference [SNR in dB] and Binaural Masking Level Difference [SNR in dB] and speech test [Oldenburger Satztest in noise [SNR in dB]. Thereby, the correlation between psycho acoustical test results and speech test results will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland